CLINICAL TRIAL: NCT00391001
Title: Taurine as an Anti-Manic Agent: A Double-Blind, Placebo-Controlled Study in Adolescents With Bipolar Disorder
Brief Title: Taurine in Adolescents With Bipolar Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Stanley Medical Research Institute (Other); Mclean Hospital (Other)
Responsible Party: Jean Frazier, MD, Cambridge Health Alliance
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHA-IRB-0131/09/05
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar Disorder
Keywords: mania; bipolar disorder; taurine; adolescents
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Taurine
- 2 (Placebo Comparator)
  Interventions: Drug: Taurine

INTERVENTIONS:
Drug: Taurine — double-blind, placebo-controlled, adjunctive medication

SUMMARY:
Recently, McLean hospital conducted a 4 month taurine study which showed a reduction in mania ratings. As a follow-up to the preliminary taurine study, and complementary to the currently ongoing double-blind, placebo-controlled trial for taurine in adults with bipolar disorder, this study will target adolescent bipolar subjects (type I) with symptoms of mania or mixed mania. To our knowledge, this would be the first study to evaluate the effects of the novel compound taurine in adolescent subjects with bipolar disorder.

We hypothesize there will be a positive response in some adolescents from taurine treatment, and this positive response will be greater than that expected by chance. This study may demonstrate that taurine is a well-tolerated and effective adjunct treatment for mania in bipolar disorder.

DETAILED DESCRIPTION:
A cohort of adolescent (ages 13-18) patients with bipolar disorder and current manic symptoms will be approached for participation in this 3-month outpatient study. Taurine or matching placebo will be administered orally, in capsules, and added to whatever medication(s) the patients are receiving from their clinicians. The specific medications and dosages will be determined solely by the subjects' non-study clinicians ("treatment-as-usual"). During the 3 months of the study, subjects will be required to keep their medications nearly constant (minor dosage adjustments for side-effects or to maintain therapeutic levels will be permitted) for the duration of the trial. Since taurine will be an adjunctive therapy, patients currently taking mood stabilizers can continue to do so. The research team will work closely with the subject and their outpatient clinician(s) to coordinate the medication issues. The results from standard rating scales for bipolar disorder research will be compared between the group receiving the taurine and the group receiving placebo.

The sample will include thirty adolescent (ages 13-18) outpatients with bipolar disorder, type I. The study will be 3 months long.

Study Drugs: The cohort will be randomized to receive either taurine or matching placebo (microcellulose). Taurine and placebo will be provided in 500 mg vegetable capsules.

Follow-up visits and clinical ratings:

During the baseline visit, a detailed psychiatric and medical history will be obtained. The adolescent will start study medicine at that time. The following standard rating scales will be performed:

1. Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Episode (K-SADS-PL) with additional mood onset and offset items derived from the WASH-U K-SADS (K-SADS-PL-W) (Kaufman 1997).
2. Young Mania Rating Scale (YMRS; 11 item structured interview; Young et al 1978).
3. Children's Depression Rating Scale - Revised (CDRS-R; Overholser 1995).
4. The ADHD Rating Scale (ARS-IV; DuPaul 1998).
5. Clinical Global Impression scale - Bipolar version (CGI-BP; Guy 1976).
6. Children's Global Assessment Scale (CGAS; Shaffer 1995).
7. Montgomery-Asberg Depression rating Scale (MADRS; Montgomery & Asberg 1979).
8. Brief Adverse Effect Rating Scale.
9. Brief Psychiatric Rating Scale for Children (BPRS-C; Overall & Pfefferbaum 1982).
10. Safety Assessment (derived from our group's ongoing treatment studies).

After the baseline evaluation, subjects will be evaluated every week for 1 month, and then every 2 weeks for the remainder of the 3 months. The same rating scales will be performed at each follow-up visit, except for the KSADS-PL-W and the ARS-IV. Instead of the full KSADS-PL-W at the follow-up visits, only the screening questions for mania and depression will be performed in order to aid in the determination of syndromic recovery or recurrence. In addition, patients will maintain a daily Mood Diary, which will be reviewed at each study visit to elicit symptom recall.

All ratings will be performed by blind study personnel, who will not know whether the patient is receiving taurine or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet DSM-IV-TR criteria for bipolar disorder (type I), and current hypomania, mania, or mixed mania.
* Subjects must be between the ages of 13 through 18 years.
* Medications ("treatment-as-usual") stable x2 weeks
* Subjects must be able to assent to their participation in the study.
* Subjects must agree to avoid taking supplemental taurine (e.g. from over-the-counter preparations, energy drinks, etc).

Exclusion Criteria:

* Co-morbid serious mental illness.
* Significant medical or neurological illness, including: seizure disorders, severe respiratory illness or cardiac conditions, known cerebrovascular disease, hypo- or hypertension, diabetes mellitus, and immune, endocrine, renal or hepatic dysfunction (the study team does not wish to enroll any subjects at increased risk for complications or who require additional clinical monitoring due to their medical illness).
* Pregnant subjects. It is not known what effects taurine supplementation would have on a fetus. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded.
* Patients who, in the investigator's judgment, pose a current serious suicidal or homicidal risk, or patients who will not likely be able to comply with the study protocol.
* Patients who meet DSM-IV-TR criteria for current substance abuse or substance dependence.
* Patients who are regularly taking supplemental taurine at the time of screening.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS; 11 item structured interview; Young et al 1978). | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Jean Frazier, MD, Principal Investigator — Cambridge Health Alliance
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Cambridge Health Alliance Child & Adolescent Neuropsychiatric Research Program, Medford, Massachusetts

REFERENCES:
- [Background] Redmond HP, Stapleton PP, Neary P, Bouchier-Hayes D. Immunonutrition: the role of taurine. Nutrition. 1998 Jul-Aug;14(7-8):599-604. doi: 10.1016/s0899-9007(98)00097-5. PMID 9684263
- [Background] Stoll AL, Severus WE, Freeman MP, Rueter S, Zboyan HA, Diamond E, Cress KK, Marangell LB. Omega 3 fatty acids in bipolar disorder: a preliminary double-blind, placebo-controlled trial. Arch Gen Psychiatry. 1999 May;56(5):407-12. doi: 10.1001/archpsyc.56.5.407. PMID 10232294
- [Background] Thornton L, Griffin E. Evaluation of a taurine containing amino acid solution in parenteral nutrition. Arch Dis Child. 1991 Jan;66(1 Spec No):21-5. doi: 10.1136/adc.66.1_spec_no.21. PMID 1899989
- [Background] Van Gelder NM, Sherwin AL, Sacks C, Anderman F. Biochemical observations following administration of taurine to patients with epilepsy. Brain Res. 1975 Aug 29;94(2):297-306. doi: 10.1016/0006-8993(75)90063-3. PMID 807299